CLINICAL TRIAL: NCT03596073
Title: A Pilot Trial of Topical Calcipotriene Treatment for Breast Cancer Immunoprevention
Brief Title: Topical Calcipotriene Treatment for Breast Cancer Immunoprevention
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Interim analysis did not show the required cytokine induction by topical calcipotriene to justify continuation of the trial
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Shadmehr Demehri, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-040
Record Dates: First submitted 2018-07-10; First posted 2018-07-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Calcipotriene Ointment (Experimental): -Topical Calcipotriene Ointment will be administered by the participants to their upper extremities twice a day for the period between core biopsy and surgical removal of their breast lesion
  Interventions: Drug: Topical Calcipotriene Ointment
- Topical Vaseline (Placebo Comparator): -Topical Vaseline will be administered by the participants to their upper extremities twice a day for the period between core biopsy and surgical removal of their breast lesion
  Interventions: Other: Topical Vaseline

INTERVENTIONS:
Drug: Topical Calcipotriene Ointment — Calcipotriene is a form of vitamin D. It works by slowing down the growth of skin cells.
  Arms: Topical Calcipotriene Ointment
Other: Topical Vaseline — Placebo
  Arms: Topical Vaseline

SUMMARY:
This research study is studying a topical ointment called calcipotriene to see if it can stimulate the immune cells against the breast lesion in ways that would prevent its recurrence after surgical removal

DETAILED DESCRIPTION:
The investigators are doing this research study to find out how topical calcipotriene ointment affect people who have breast cancer, and what impact that may have on those who are at risk of developing breast cancer in the future. The investigators hope that what they learn will lead to the development of a new medication for the treatment and prevention of breast cancer.

Abnormal breast lesions can be benign, premalignant or malignant. These lesions are being targeted by the topical calcipotriene ointment. The investigators aim to determine whether this topical treatment can stimulate the immune cells against the breast lesion in ways that would prevent its recurrence after surgical removal.

Calcipotriene ointment is approved by the U.S. Food and Drug Administration (FDA) to treat psoriasis, but calcipotriene ointment is not approved by the FDA to treat breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed benign, premalignant or early malignant breast lesions on core biopsy that will proceed directly to surgical removal without any intervening neoadjuvant chemotherapy.
* Patients diagnosed with benign breast lesions (papilloma and sclerosing lesion), flat epithelial atypia, atypical ductal hyperplasia, lobular carcinoma in situ (Tis N0 M0; stage 0), ductal carcinoma in situ (Tis N0 M0; stage 0), primary invasive ductal and lobular carcinoma (T1or2 N0or1 M0; stage I-II), who will directly receive surgery and no neoadjuvant chemotherapy.
* Patients with hormone receptor positive, Her2 positive and triple negative cancers will be eligible.
* Patients with multicentric and multifocal tumors will be eligible.
* Age 45 years. To avoid the impact of menstrual cycles-associated alterations in the immune environment of the breast, the age is limited to post-menopausal women.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants scheduled to undergo neoadjuvant therapy for breast cancer.
* Participants with metastatic breast cancer.
* Participants with history of breast cancer in the past 5 years.
* Participants with immunosuppression (e.g., organ transplant recipients and patients with autoimmune diseases requiring immunosuppressive medications including >5mg daily prednisone, methotrexate, cyclosporine, azothioprine, tacrolimus and TNFα blocking agents)
* Participants with the history of hypercalcemia or clinical evidence of vitamin D toxicity.
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to topical calcipotriene ointment.
* Pregnant women are excluded from this study because topical calcipotriol ointment is a category C agent and its impact on developing fetus is unknown. In addition, premenopausal women are excluded from this study due to the impact of menstrual cycles on immune environment of the breast.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The changes in the magnitude of CD3+ T cell infiltration in tumor microenvironment | 3 Weeks
  The change in the number of CD3+ T cells per high power microscope field in tumor microenvironment from the time of initial needle core biopsy to surgical excision.

SECONDARY OUTCOMES:
The comprehensive changes in tumor immune microenvironment | 3 Weeks
The changes in tumor immune microenvironment in patients with neoplastic tumors versus benign lesions | 3 Weeks
The changes in tumor immune microenvironment in patients with stage I-II, versus stage 0 tumors | 3 Weeks
The changes in tumor immune microenvironment in patients with hormone receptor and Her2 positive versus triple negative tumors | 3 Weeks
Serum Serum Thymic Stromal Lymphopoietin (TSLP) levels (picogram/milliliter) before and after topical calcipotriene treatment compared to Vaseline control group | 3 Weeks
Disease free survival | From the start of treatment up to 15 years
  The duration of time measured from the start of treatment until the time of disease progression or death, whichever occurs first.
Number of Participants with Treatment Related Adverse Events | From the start of treatment until 30 days after the end of treatment, up to 2 months
  Adverse events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE v4).

CONTACTS AND LOCATIONS:
Overall Officials: Shadmehr Demehri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No